CLINICAL TRIAL: NCT06271031
Title: Computer Simulation Model of Patients With Bloodstream Infection, Sepsis and Systemic Infection (CSM-BSI)
Brief Title: Process Mapping and Data Collection to Inform a Computer Simulation Model of Hospitalised Patients With Bloodstream Infection, Sepsis and Systemic Infection
Acronym: CSM-BSI
Status: Recruiting | Type: Observational
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: LHS0211
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-10

CONDITIONS: Sepsis; Bloodstream Infection; Bacteraemia
MeSH Terms: conditions — Sepsis; Toxemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to create a computer simulation of patients with bloodstream infection to understand how changes in healthcare policies and resources affect patient treatment. This simulation will help doctors and health-care decision makers make better choices in treating these patients and avoid overusing antibiotics that can lead to antibiotic resistance. Antibiotic resistance is when bacteria can't be killed by antibiotics anymore. Participants will not receive treatments as this is an observational study, but the study will involve:

* Interviews with healthcare staff to understand patient care pathways.
* Analysis of historical data on bacteria causing infections and antibiotic treatments.
* A 30-day observational study to observe patient treatment for bloodstream infections.

DETAILED DESCRIPTION:
The main aim of this research is to create a computer simulation of patients with bloodstream infection. Bloodstream infection is often a severe infection (blood poisoning) that can lead to sepsis, which is a significant global health concern, causing around 66,096 deaths each year in the United Kingdom alone. Doctors and healthcare decision-makers have to make difficult decisions that balance the effective treatment of patients with sepsis and avoid the overuse of broad-spectrum antibiotics, which can lead to antibiotic resistance. By generating a virtual environment to test out different scenarios, this computer simulation model will provide insight into the projected effects of changes to hospital policy, changes in hospital resources (such as staff) and the impact of laboratory diagnostic tests. Proposed changes can be simulated in this virtual environment prior to implementation in the real healthcare system.

This study will be carried out in three parts. First, there will be interviews with healthcare staff over six months to comprehensively describe the patient pathways involved in management of bloodstream infection. Next, the project will analyse historical pseudonymised data from Liverpool University Hospitals NHS Foundation and Liverpool Clinical Laboratories to inform the characteristics of the model (in particular on the bacteria causing infections, the antibiotic treatments used, and the time it takes for patients to be treated). Finally, there will be a 30-day observational study where researchers observe the treatment of patients with bloodstream infection (without intervening or recording identifying details) to ensure that the computer model captures all the important steps involved in patient management.

ELIGIBILITY:
Inclusion Criteria:

Sub-study 2 (retrospective data collection)

* Patients who were managed within a LUFT acute hospital site (Aintree or Royal) and had a concurrent blood culture investigation requested
* Age ≥ 18 years at the time of the study. Sub-study 3 (observational study)
* Patients with blood culture investigation requested during the observation period, and staff caring for the patients.

Exclusion Criteria:

* Age < 18 years at the time of the study
* Blood culture requested but patient not managed on an acute hospital site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with presumed bloodstream infection/sepsis/systemic infection.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Generation of a software simulation model that is fine tuned to the observed data. | 2 years
  The main outcome is the generation of a software simulation model that is calibrated to the observed data. The study team consists of individuals with experience in model construction and calibration.

SECONDARY OUTCOMES:
Exploration of the performance of the model in different hypothesised scenarios. | 6 months
  Secondary outcomes of this study are the exploration of the performance of the model in different hypothesised scenarios. The scenarios and outcome metrics are dependant on the final model delivered, but as an example may include the following: Time from presentation to hospital to time to administration of antibiotics active against the infecting pathogen in a simulated model which includes a novel diagnostic test for antimicrobial resistance, vs a model that does not include one.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro D Gerada, Principal Investigator — University of Liverpool
Locations (1):
- Liverpool University Hospitals Foundation Trust, Liverpool, United Kingdom

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT06271031/Prot_ICF_000.pdf